CLINICAL TRIAL: NCT06556602
Title: Methadone Patient Access to Collaborative Treatment (MPACT)
Brief Title: Methadone Patient Access to Collaborative Treatment
Acronym: MPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 456483
Record Dates: First submitted 2024-07-16; First posted 2024-08-16 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Opioid Use Disorder; Staff; Patients
Keywords: Methadone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1, 18-month simultaneous cluster randomized controlled trial in 30 clinics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPACT Intervention (Experimental): Enrolled clinic staff will be exposed to the MPACT intervention components over the trial period. This includes accredited training, clinic self assessment, reflective supervision for counseling/peer/case management staff, and wellness education with navigation to trauma symptoms assessment and resources including trauma treatment. Periodic surveys of staff and patients will be conducted to assess outcome measures (primary and secondary) and patient chart reviews will verify patient outcomes.
  Interventions: Other: MPACT
- Control for MPACT (No Intervention): Enrolled clinic staff will not receive any portion of the intervention. Periodic surveys of staff and patients will be conducted to assess outcome measures (primary and secondary) and patient chart reviews will verify patient outcomes.

INTERVENTIONS:
Other: MPACT — Four components are part of this intervention: 1) accredited training about patient centered, trauma-informed care and the standard of care under the current federal regulation (42CFRpart8), 2) education about trauma and trauma symptoms including vicarious (work related) trauma and navigation to symptoms screening and resources including treatment, 3) reflective supervision for counseling, case management and peer staff, and 4) clinic self assessment for trauma-informed and patient centered care
  Arms: MPACT Intervention

SUMMARY:
The trial of Methadone Patient Access to Collaborative Treatment (MPACT) will establish the impact of the intervention on patient outcomes of methadone treatment retention and in treatment overdose.

It will also establish the impact of patient and staff trauma symptoms and clinic practice change on MPACT intervention implementation.

DETAILED DESCRIPTION:
This MPACT trial will involve finalizing the refined MPACT intervention (materials, training) and conducting a Hybrid Type 1, 15-month cluster randomized controlled trial in 30 clinics with 600 patients (20/clinic) and 480 staff (18/clinic) to assess MPACT effect on patient outcomes and examine the relationship between staff trauma outcomes and MPACT implementation. R33 Specific AIMS:

AIM 1: Quantify the effects of MPACT on methadone treatment (MMT) practice change and opioid treatment program (OTP) culture.

AIM 2: Determine the efficacy of MPACT on MMT retention, in-MMT overdose and patient and staff post traumatic stress symptoms (PTSS) outcomes.

AIM 3: Evaluate the effect of patient and staff trauma symptoms on primary outcomes and staff MPACT implementation.

ELIGIBILITY:
Inclusion Criteria:

* Staff providing methadone treatment services at the enrolled opioid treatment programs

Exclusion Criteria:

* Patients receiving methadone treatment at the enrolled opioid treatment programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Days in Treatment to treatment interruption | 18 months
  Time (days) to treatment interruption
Time to treatment cessation | 18 months
  Time to treatment cessation (tolerance of 30 days)
In Treatment- Point in time | 18 months
  Point in time in treatment (0 day, 30 day, 60, day, 90 day)
Number of patients reporting opioid overdoses while in methadone treatment | 18 months
  Reported overdoses by patients in methadone treatment during the trial period by survey measured at 5 points during the study period.

SECONDARY OUTCOMES:
Number of staff experiencing vicarious (work related) stress | 18 months
  Post traumatic stress symptoms and vicarious (work related) trauma symptoms measured by the Vicarious Trauma Scale (VTS). Total scores can be grouped into three categories to represent low (8-28), moderate (29-42) and high (43-56) levels of vicarious trauma symptoms
Number of patients and staff experiencing post traumatic stress symptoms | 18 months
  Post traumatic stress symptoms measured by the 8-item PCL-5 measuring post traumatic stress symptoms. Scores range from 0-80, with higher scores representing greater levels of traumatic stress symptomatology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona College of Medicine, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
A Data Management and Sharing Plan has been filed with the National Institute on Drug Abuse.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within 2 years of study completion
Access Criteria: See Data Management and Sharing Plan

REFERENCES:
- [Derived] Meyerson BE, Davis A, Crosby RA, Linde-Krieger LB, Brady BR, Carter GA, Mahoney AN, Frank D, Rothers J, Coffee Z, Deuble E, Ebert J, Jablonsky MF, Juarez M, Lee B, Lorenz HM, Pava MD, Tinsely K, Yousaf S. Methadone Patient Access to Collaborative Treatment: Protocol for a Pilot and a Randomized Controlled Trial to Establish Feasibility of Adoption and Impact on Methadone Treatment Delivery and Patient Outcomes. JMIR Res Protoc. 2025 Apr 15;14:e69829. doi: 10.2196/69829. PMID 40105313